CLINICAL TRIAL: NCT00511680
Title: Treating Depression in African American Elders: A Community-Academic Partnership
Brief Title: Beat the Blues: Treating Depression in African American Elders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Laura N. Gitlin, Director, Center for Innovative Care in Aging, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 1R01MH079814 (NIH)
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Depression; Stress Reduction; Behavioral Activation Treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral based In-home Intervention (Experimental): This group will recieve up to 10 1-hour sessions over a 4 month period.
  Interventions: Behavioral: Behavioral Based In-Home Intervention

INTERVENTIONS:
Behavioral: Behavioral Based In-Home Intervention — The 10 session intervention delivered by a social worker in the home includes five treatment components (education, referral, care management, stress reduction, behavioral activation). Each component has been shown to be effective in treating depression in previous research.

SUMMARY:
The specific primary aims of the study are to:

1. Test the immediate effect of the intervention at 4-months on depression in urban African American older adults (primary trial outcome; between group comparison). Hypothesis: Participants in the intervention group will report fewer depressive symptoms in comparison to control group participants receiving usual care.
2. Test the maintenance effect of the intervention at 8-months on depression (within group comparison). Hypothesis: Participants in the intervention group will maintain reduced symptom presentation from 4 to 8 months.
3. Evaluate acceptability (social validity) of the intervention and extent of engagement in activities by study participants (both intervention and wait-list control subjects).

A secondary aim of this study is to assess the feasibility of conducting a clinical trial embedded in a community service setting and its dissemination using a community-academic partnership. We also propose three exploratory aims. First, we seek to evaluate the mechanisms of action, or pathways, by which treatment gains are obtained (Gitlin et al., 2000). Given that behavioral activation represents conceptually the key active ingredient of the proposed intervention, we plan to evaluate its mediational effect. Second, we seek to evaluate whether the intervention has a differential treatment effect based on a study participant's gender, age, and living arrangement (alone or with others). Given that previous research suggests that participant characteristics may moderate depressive symptoms and treatment outcomes, these exploratory analyses will provide insight as to whether this particular treatment benefits some groups more than others. Third, we seek to evaluate whether the intervention has short and long-term effects on quality of life, functional difficulty, and self-efficacy to manage day-to-day tasks. Previous research has shown that depressive symptoms exacerbate functional decline such that minimizing distress may have the added value of enhancing function and perceived efficacy for this group over time.

ELIGIBILITY:
Inclusion Criteria:

* African American
* ≥55 years of age
* English speaking
* Cognitively intact (MMSE >24)
* Depressed as measured by a score ≥5 on the PHQ-9
* Must have a telephone
* Planning to live in the area for 8 months

Exclusion Criteria:

* Not African American
* <55 years of age
* Does not speak English
* MMSE<24
* Not depressed as measures by a score of <5 on the PHQ-9
* Does not have a telephone
* Does not plan to live in the area for 8 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline, t2, t3

CONTACTS AND LOCATIONS:
Overall Officials: Laura N. Gitlin, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gitlin LN, Harris LF, McCoy MC, Hess E, Hauck WW. Delivery Characteristics, Acceptability, and Depression Outcomes of a Home-based Depression Intervention for Older African Americans: The Get Busy Get Better Program. Gerontologist. 2016 Oct;56(5):956-65. doi: 10.1093/geront/gnv117. Epub 2015 Nov 25. PMID 26608333
- [Derived] Gitlin LN, Szanton SL, Huang J, Roth DL. Factors mediating the effects of a depression intervention on functional disability in older African Americans. J Am Geriatr Soc. 2014 Dec;62(12):2280-7. doi: 10.1111/jgs.13156. PMID 25516024
- [Derived] Gitlin LN, Roth DL, Huang J. Mediators of the impact of a home-based intervention (beat the blues) on depressive symptoms among older African Americans. Psychol Aging. 2014 Sep;29(3):601-11. doi: 10.1037/a0036784. PMID 25244479
- [Derived] Gitlin LN, Harris LF, McCoy MC, Chernett NL, Pizzi LT, Jutkowitz E, Hess E, Hauck WW. A home-based intervention to reduce depressive symptoms and improve quality of life in older African Americans: a randomized trial. Ann Intern Med. 2013 Aug 20;159(4):243-52. doi: 10.7326/0003-4819-159-4-201308200-00005. PMID 24026257
- [Derived] Jutkowitz E, Pizzi L, Hess E, Suh DC, Gitlin LN. Comparison of three societally derived health-state classification values among older African Americans with depressive symptoms. Qual Life Res. 2013 Aug;22(6):1491-8. doi: 10.1007/s11136-012-0263-y. Epub 2012 Sep 13. PMID 22972437
- [Derived] Gitlin LN, Harris LF, McCoy M, Chernett NL, Jutkowitz E, Pizzi LT; Beat the Blues Team. A community-integrated home based depression intervention for older African Americans: [corrected] description of the Beat the Blues randomized trial and intervention costs. BMC Geriatr. 2012 Feb 10;12:4. doi: 10.1186/1471-2318-12-4. PMID 22325065